CLINICAL TRIAL: NCT03917251
Title: The Effects of Trans Venous Cardiac Pacing on Coronary Microvascular Function and Hemodynamics
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: PI left the institution
Sponsor: University of Nebraska (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Basic Science
Other Study IDs: 0898-18-FB
Record Dates: First submitted 2019-03-03; First posted 2019-04-17 (Actual); Last update posted 2024-09-03 (Actual); Status verified 2024-08

CONDITIONS: Coronary Microvascular Disease; Cardiac Pacemaker Syndrome
Keywords: coronary microvascular dysfunction
MeSH Terms: conditions — Microvascular Angina

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Right ventricular Pacemaker (Other): Patients with right ventricular pacing and evidence of coronary ischemia who have evidence of coronary ischemia who are to undergo coronary angiogram.When an intermediate stenosis (40-80%) has been identified angiographically, this lesion will undergo further hemodynamic assessment, All data including resting flow, FFR, CFR, vital signs, arrhythmias and patient symptoms will be recorded twice: once when the pacemaker is programmed to pace, and once when the PPM is reprogrammed such that the pacemaker is no longer pacing.
  Interventions: Diagnostic Test: Coronary flow and pressure measurement in patients with ventricular pacing
- Biventricular Pacemaker (Other): Patients with Biventricular pacing and evidence of coronary ischemia who have evidence of coronary ischemia who are to undergo coronary angiogram.When an intermediate stenosis (40-80%) has been identified angiographically, this lesion will undergo further hemodynamic assessment, All data including resting flow, FFR, CFR, vital signs, arrhythmias and patient symptoms will be recorded twice: once when the pacemaker is programmed to pace, and once when the PPM is reprogrammed such that the pacemaker is no longer pacing.
  Interventions: Diagnostic Test: Coronary flow and pressure measurement in patients with ventricular pacing

INTERVENTIONS:
Diagnostic Test: Coronary flow and pressure measurement in patients with ventricular pacing — Coronary flow and pressure measurement in patients with ventricular pacing

SUMMARY:
The study will examine role of transvenous pacing on coronary microcirculation.

DETAILED DESCRIPTION:
To study the role of transvenous pacing on the coronary microcirculation. This will be accomplished by gathering data from invasive Fractional Flow Reserve (FFR) and Coronary Flow Reserve (CFR) with and without ventricular pacing.

ELIGIBILITY:
Inclusion Criteria:

All patients 19 years of age or older with clinical evidence of coronary ischemia undergoing coronary angiogram, and who have a pacemaker.

Exclusion Criteria:

* Acute ST segment myocardial infarction
* Known sensitivity or contraindication to the agents planned for administration during coronary angiography
* Pacemaker dependent patients
* Pregnancy
* Hypotension (a systolic blood pressure lower than 90mmHg) that would preclude the administration of adenosine
* Severe renal dysfunction, defined as a estimated glomerular filtration (eGFR) less than 30ml/min, confirmed by recent testing
* Study subject has any underlying disorder that, in the opinion of the investigator, precludes them from giving informed consent at the time of enrollment

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-10-07 (Estimated); Primary Completion 2021-10-07 (Actual); Study Completion 2021-10-07 (Actual)

PRIMARY OUTCOMES:
Patients that exhibit coronary microvascular resistance and dysfunction as reflected by FFR | Up to 12 months
  Microvascular dysfunction with pacing

SECONDARY OUTCOMES:
Patients that exhibit coronary microvascular resistance and dysfunction as reflected by CFR | Up to 12 months
  Microvascular dysfunction with pacing

CONTACTS AND LOCATIONS:
Overall Officials: Nashwa Abdulsalam, MD, Principal Investigator — University of Nebraska

IPD SHARING:
Plan to Share IPD: No